CLINICAL TRIAL: NCT02511392
Title: Repetitive Transcranial Magnetic Stimulation in the Treatment of Obsessive-Compulsive Disorders: Double Blind Randomized Clinical Trial
Brief Title: Repetitive Transcranial Magnetic Stimulation in the Treatment of Obsessive Compulsive Disorders
Acronym: rTMS-OCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman M. Khedr, Clinical professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: rTMS-OCD
Record Dates: First submitted 2015-07-28; First posted 2015-07-30 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Obsessive Compulsive Disorders
MeSH Terms: conditions — Compulsive Personality Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1: Real rTMS-1 Hz (Active Comparator): Included 15 patients, they received 1 Hz rTMS with intensity of 100% of the RMT continuous with total 2000 applied in 200 trains, each of 10 pulses, with 5 seconds intertrain interval
  Interventions: Procedure: rTMS-1Hz
- Group 2: Real rTMS-10 Hz (Active Comparator): Included 15 patients, they received 10 Hz rTMS with intensity of 100% of the RMT applied in 10 trains, each of them 200 pulses, with 20 seconds intertrain interval
  Interventions: Procedure: rTMS-10 Hz
- Group 3: Sham rTMS (Sham Comparator): Included 15 patients; they received the same number of pulses 2000 pulse applied in 200 trains, each of 10 pulses, with 5 seconds intertrain interval, but coil was placed over the same area but perpendicular to the scalp.
  Interventions: Procedure: Sham rTMS

INTERVENTIONS:
Procedure: rTMS-1Hz
  Arms: Group 1: Real rTMS-1 Hz
Procedure: rTMS-10 Hz
  Arms: Group 2: Real rTMS-10 Hz
Procedure: Sham rTMS
  Arms: Group 3: Sham rTMS

SUMMARY:
Objectives.-Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive stimulation methods that became widely used as therapeutic tools in neuropsychiatric research. The aim of this study is to Evaluate the therapeutic impact of different frequencies of repetitive transcranial stimulation (1HZ, 10HZ) in OCD patients. Material and Methods; Forty five patients of OCD were participated in the study. All patients fulfilled the diagnostic criteria of DSM-IV-TR. The mean age of the patients was 27.1+4.5 years. Each patient was subjected to the following: Yale-Brown obsessive compulsive scale (Y-BOCS), Hamilton Anxiety Rating Scale (HAM-A), and Clinical Global Impression - Severity scale (CGI-S). The patients were randomly classified into three equal groups using closed envelop: 1st group received 1 Hz rTMS at 100% of the RMT, 2nd group received 10 Hz rTMS with intensity of 100% of the RMT and 3rd group was sham group received the sham stimulation with a total 2000 pulses every day for each group for 10 sessions. Follow up of the patients using the same previous scales after the end of sessions and 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* All patients fulfilled the diagnostic criteria of DSM-IV-TR

Exclusion Criteria:

* Patients with comorbid psychiatric disorder .

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
changes of Y-BOCS | Base line and after 3 months
  Yale-Brown obsessive compulsive scale (Y-BOCS). It is an observer-rated scale that measures the severity of OCD symptoms. It is not a diagnostic tool. It is formed of 2 subscales, one for obsessions and another for compulsions. Each subscale consists of 5 items; і) time spent in the symptoms, іі) interference from the symptoms, ііі) subjective distress from symptoms, іv) resistance over symptoms, v) control over symptom. Each of these is rated from 0 (no symptoms) to 4 (extreme symptoms). The total Y-BOCS score ranges between: 0-7 subclinical 8-15 mild 16-23 moderate 24-31 severe 32-40 extreme (Goodman et al., 1989).

SECONDARY OUTCOMES:
Changes in HAM-A score | Base line and after 3 months
  Hamilton Anxiety Rating Scale (HAM-A). The HAM-A was one of the first rating scales developed to measure the severity of anxiety symptoms by Max Hamilton (1959), and is still widely used today in both clinical and research settings. The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where 0-14,normal range; 15-28, mild to moderate anxiety; 29-42, severe anxiety; 43-56, very severe anxiety. The scale has been translated into Arabic by Lotfy Fatem (1994).
Changes in CGI-S score | Base line and after 3 months
  Clinical Global Impression - Severity scale (CGI-S): It is a 7- point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. (Guy 1976). Considering total clinical experience, a patient is assessed on severity of mental illness at the time of rating 1,normal,not at all ill; 2,borderline mentally ill; 3,mildly ill; 4,moderately ill; 5,markedly ill; 6,severely ill; or 7, extremely ill. (Rush 2000).